CLINICAL TRIAL: NCT01015729
Title: An Open-Label, Randomized, Single-Center, 3-Way Crossover Study Comparing The Therapeutic Efficacy of a Fixed Dose Combination Capsule of Esomeprazole 20 mg And Acetylsalicylic Acid (ASA) 81 mg With Free Combinations of ASA Tablet 81 mg And Esomeprazole 20 mg as a Capsule or Tablet in Patients At Risk of Gastrointestinal Events Using Low Dose ASA for Cardiovascular Protection
Brief Title: Study Comparing Esomeprazole and ASA Combined Together as One Capsule Versus These Medications Taken Separately
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D961FC00008
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Peptic Ulcer Disease
Keywords: Bioequivalence; ASA; Esomeprazole; peptic ulcer disease; pH measurements
MeSH Terms: conditions — Peptic Ulcer | interventions — Esomeprazole; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Esomeprazole 20 mg/ASA 81 mg Fixed Dose Combination Capsule
  Interventions: Drug: Esomeprazole/ASA Fixed Combination
- 2 (Active Comparator): Esomeprazole Clinical Trial Capsule 20 mg and 1 Aspirin® Non Enteric Coated Immediate Release Tablet 325 mg
  Interventions: Drug: Esomeprazole; Drug: ASA
- 3 (Active Comparator): Esomeprazole MUPS Tablet 20 mg and 1 Aspirin® Non Enteric Coated Immediate Release Tablet 325 mg
  Interventions: Drug: Esomeprazole; Drug: ASA

INTERVENTIONS:
Drug: Esomeprazole/ASA Fixed Combination — Capsule, oral, single dose
  Arms: 1
Drug: Esomeprazole — oral, single dose
  Other Names: Nexium
  Arms: 2; 3
Drug: ASA — Tablet, oral, single dose
  Other Names: Aspirin
  Arms: 2; 3

SUMMARY:
The purpose of this study is to investigate whether a fixed dose combination (FDC) capsule of esomeprazole 20 mg and acetylsalicylic acid (ASA) 81 mg has equivalent therapeutic efficacy compared to each of 2 free combinations of ASA tablet 81 mg plus esomeprazole 20 mg in patients at risk of gastrointestinal events using low dose ASA for cardiovascular protection.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male and female subjects, aged 18 years or older with a documented history of uncomplicated peptic ulcer(s), or aged 65 years or older
* Body Mass Index (BMI = weight/height2) greater than or equal to 18.5 kg/m2 and less than or equal to 35.0 kg/m2

Exclusion Criteria:

* Known history of hypersensitivity to esomeprazole (e.g. Nexium®) or related drugs such as omeprazole (e.g. Losec®, Prilosec®), lansoprazole (e.g. Prevacid®, Hp-PAC®), pantoprazole (e.g. Pantoloc®, PANTO® IV), or rabeprazole (e.g. Pariet™), a known hypersensitivity to ASA (e.g. Aspirin®) and/or related drugs such as ibuprofen (e.g. Motrin®, Advil®), indomethacin (e.g. Indocin®), diclofenac (e.g. Voltaren®), naproxen (e.g. Aleve®, Naprosyn®), or ketoprofen (e.g. Rhovail®).
* Significant history of pulmonary, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, or gastrointestinal disease (with the exception of uncomplicated peptic ulcer), unless deemed NCS by the Principal Investigator or Sub-investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time that intragastric pH is maintained > 4.0 during the 24-hour recording period | pH is measured over a 24-hour period following dosing on Day 5 after repeated oral administartion/dosing

SECONDARY OUTCOMES:
Percentage of time that intragastric pH is maintained > 3.0 during the 24-hour recording period | pH is measured over a 24-hour period following dosing on Day 5 after repeated oral administartion/dosing
Median 24-hour intragastric pH | pH is measured over a 24-hour period following dosing on Day 5 after repeated oral administartion/dosing
Gastrointestinal symptom (Global Overall Symptoms questionnaire) | GOS questionnaire will be adminsited on day 5

CONTACTS AND LOCATIONS:
Overall Officials: TJorgen Nasdal, MD, PhD, Study Director — AstraZeneca R&D; Pierre Geoffroy, M.D. C.M., M.Sc., F.C.F.P., Principal Investigator — Biovail Contract Research (BCR)
Locations (1):
- Research Site, Scarborough Village, Ontario, Canada